CLINICAL TRIAL: NCT04694183
Title: PD-1 Inhibitor Plus Chemotherapy as Conversion Therapy in Unresectable Gastric Cancer (STARS-GC01): A Single-arm, Single-center, Prospective Clinical Study.
Brief Title: The Conversion Therapy of Chemotherapy Plus Camrelizumab in Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quan Wang (Other)
Responsible Party: Sponsor-Investigator, Quan Wang, Doctor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARS-GC01
Record Dates: First submitted 2020-11-20; First posted 2021-01-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Stomach Neoplasms
Keywords: gastric cancer; metastasis; conversion therapy; immune checkpoint inhibitors; camrelizumab
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — camrelizumab; S 1 (combination); Oxaliplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversion therapy (Experimental): Camrelizumab combined with chemotherapy selected per metastasis site.
  Interventions: Drug: Camrelizumab; Drug: S-1; Drug: Oxaliplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — 200mg, intravenous drip administration, d1, every 3 weeks.
  Other Names: SHR-1210
Drug: S-1 — Oral, d1-14, every 3 weeks.
  Other Names: Tegafur Gimeracil Oteracil Potassium Capsule
Drug: Oxaliplatin — 130mg/m² intravenous drip administration, d1, every 3 weeks(For patients with liver and/or para-aortic lymph node metastasis).
Drug: Paclitaxel — Intraperitoneal paclitaxel 20 mg/m² and intravenous paclitaxel 50 mg/m² on days 1 and 8, every 3 weeks(For patients with peritoneal metastasis ).

SUMMARY:
Gastric cancer is one of the most common malignant tumors of the digestive tract. Gastric cancer patients diagnosed for the first time in China have a higher proportion of advanced stages and a higher postoperative metastasis rate.Studies have shown that patients with good pathological response after preoperative neoadjuvant therapy (such as tumor regression grade, TRG0 or 1) have a better prognosis.The purpose of this study is to treat patients with advanced gastric cancer who are difficult to perform R0 surgery with chemotherapy combined with immunotherapy. At the same time as the primary cancerous lesions are reduced, the distant metastatic lesions are effectively controlled in order to perform R0 surgery and to improve the survival rate of patients with advanced gastric cancer.

DETAILED DESCRIPTION:
The interventions include camrelizumab and chemotherapy selected based on the use of different metastatic sites as conversion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates in the study with full informed consent and signs a written informed consent form.
2. Age 18-75 years old, male or female.
3. HER-2 negative unresectable gastric cancer.
4. Patients with gastric cancer who PD-L1+（CPS≥1）or MSI-H/dMMR, or EBV（+）.
5. Patients were assessed by physicians before enrollment to determine eligibility for conversion therapy.
6. The expected survival time of the patient is≥ 12 weeks.
7. ECOG 0-1.
8. The patient has good organ function: no blood transfusion or colony-stimulating factor and thrombopoietin have been received in the 14 days before the first study, neutrophil count ≥1.5×109/L, platelet count ≥80×109/ L hemoglobin ≥ 80 g/L, serum creatinine ≤ 1.5 times the upper limit of normal (ULN), total bilirubin ≤ 1.5 times the upper limit of normal (ULN), ALT, AST ≤ 2.5 times ULN (without liver metastasis) or ≤ 5 times ULN (such as liver metastasis occurred), albumin ≥30 g/L. Requirements for coagulation function: International normalized ratio (INR) ≤ 1.5 times ULN, prothrombin time (PT) ≤ 1.5 times ULN, activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN. Requirements for electrolytes: the corrected serum calcium, blood potassium, and blood magnesium are within the normal range;
9. Women of childbearing age are required to have a pregnancy test (serum or urine) within 7 days of entry and the results are negative and are willing to use appropriate methods of contraception during the trial and 8 weeks after the last drug is given. For men, it should be surgical sterilization or consent to the use of appropriate methods of contraception during the trial and 8 weeks after the last administration of the experimental drug.

Exclusion Criteria:

1. Those who are known to be allergic to the study drug or any of its excipients or have had severe allergic reactions.
2. Patients who have received chemotherapy and monoclonal antibodies within 21 days and those who have received radiotherapy within 14 days.
3. Participated in other clinical trials within 21 days before screening.
4. Other malignant tumors have been diagnosed within 5 years before entering the study, except for skin basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or intraductal carcinoma in situ of the breast that can be treated locally and cured.
5. There is uncontrollable or symptomatic active central nervous system (CNS) metastasis, which can be manifested as clinical symptoms, cerebral edema, spinal cord compression, cancerous meningitis, leptomeningeal disease and/or progressive growth; imaging Prompt asymptomatic spinal cord compression, except for those who have been evaluated by specialists as stable and do not need treatment for the time being; For those who have received CNS metastasis treatment, imaging examinations during the screening period have shown that they have been stable for ≥4 weeks and have been stopped before the first study administration Except for systemic hormone therapy (prednisone or other curative hormones with a dose> 10 mg/day) for ≥ 4 weeks.
6. Poorly controlled pleural effusion, abdominal effusion, or pericardial effusion.
7. Poorly controlled tumor-related pain; patients who need analgesic treatment, must receive a stable dose of treatment before participating in the study; should be suitable for palliative radiotherapy (for example, bone metastasis or metastasis that causes nerve damage) before enrollment. If appropriate, consider local treatment of asymptomatic metastatic lesions whose further growth may cause functional defects or intractable pain (for example, epidural metastases not related to spinal cord compression).
8. Peripheral neuropathy or hearing loss ≥ 2 (according to NCI-CTCAE 5.0).
9. Pregnant or (confirmed by blood or urine HCG test) or breastfeeding women or subjects of childbearing age are unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until after the last trial treatment at least 6 months.
10. Patients with moderate to severe liver and kidney dysfunction.
11. Diabetes that is difficult to control (refers to the large fluctuations in blood glucose under standard insulin treatment and frequent blood glucose monitoring, which affects the life of the patient and frequent hypotension).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | Within 1 month of surgery.
  Defined as no residue under the microscope after resection

SECONDARY OUTCOMES:
Pathologic complete response | Within 1 month of surgery.
  The number of people who have achieved complete pathological remission accounted for the proportion of people who met the plan.
Overall survival | From the start of system therapy to death from any cause.
  The time from the start of system therapy to the death of any cause.
2-year survival rate | 2 years from the start of system therapy.
  Percentage of subjects who are alive without death event at two years.
Adverse events(all grades） | From the start of system therapy to 6 months after surgery.
  Assessed per Common Terminology Criteria for Adverse Events(CTCAE) version 5.0
Serious adverse events(≥grade 3） | From the start of system therapy to 6 months after surgery.
  Assessed per Common Terminology Criteria for Adverse Events(CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Quan Quan, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No